CLINICAL TRIAL: NCT00751322
Title: Project 2 (Mayo): Transfusion-Induced Alterations of Pulmonary and Immune Function in Mechanically Ventilated Patients
Brief Title: Transfusion-Induced Alterations of Pulmonary and Immune Function in Mechanically Ventilated Patients
Acronym: TRALI2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ognjen Gajic, Ognjen Gajic, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 07-008069; P50HL081027 (NIH)
Record Dates: First submitted 2008-09-09; First posted 2008-09-11 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Pulmonary Edemas; Blood Protein Disorders
Keywords: Pulmonary; Protein
MeSH Terms: conditions — Pulmonary Edema; Blood Protein Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): RBC transfusion of 5 days or less storage age
  Interventions: Other: RBC transfusion of 5 days or less storage age
- 2 (Active Comparator): RBC transfusion of conventional storage age
  Interventions: Other: RBC transfusion of conventional storage age

INTERVENTIONS:
Other: RBC transfusion of 5 days or less storage age — RBC transfusion of 5 days or less storage age
  Other Names: RBC
  Arms: 1
Other: RBC transfusion of conventional storage age — RBC transfusion of conventional storage age
  Other Names: RBC
  Arms: 2

SUMMARY:
Specific aim: To test whether transfusion of leukoreduced red cells of lesser storage time (versus conventional storage time) reduces mild alterations in pulmonary function and immune activation in critically ill patients with mechanically ventilated lungs.

We propose to perform a prospective, randomized, double-blind clinical trial in critically ill patients whose lungs are mechanically ventilated, and who have orders to receive transfusion of at least one unit of packed red cells, comparing pulmonary function between patients randomly allocated to receive a unit of red cells stored for 5 days or less, with similar patients randomly allocated to receive a unit of red cells stored conventionally (median 21 days). We will test the hypothesis that transfusion of red cells of lesser storage age, (5 days or less) will produce the less changes of pulmonary function and immune activation than will transfusion of red cells of conventional storage age (median 21 days).

DETAILED DESCRIPTION:
Specific aim: To test whether transfusion of leukoreduced red cells of lesser storage time (versus conventional storage time) reduces mild alterations in pulmonary function and immune activation in critically ill patients with mechanically ventilated lungs.

ELIGIBILITY:
Inclusion Criteria:

* Patients, male or female, any race or ethnicity, age 18 years or older, in one of the seven adult critical care units of the Mayo Clinic, Rochester, with mechanically ventilated lungs, requiring elective transfusion of at least one unit of red cells

Exclusion Criteria:

* transfusion of any blood component within the previous 2 hours, emergency transfusion or hemodynamic instability defined by other than a stable dose of vasoactive medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-08; Primary Completion 2010-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
We will test the hypothesis that the transfusion of red cells of lesser storage age, (5 days or less) will produce less changes of pulmonary function and immune activation than will transfusion of red cells of conventional storage age (median 21 days). | At the end of the transfusion as compared to the beginning of the transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Ognjen Gajic, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Kor DJ, Kashyap R, Weiskopf RB, Wilson GA, van Buskirk CM, Winters JL, Malinchoc M, Hubmayr RD, Gajic O. Fresh red blood cell transfusion and short-term pulmonary, immunologic, and coagulation status: a randomized clinical trial. Am J Respir Crit Care Med. 2012 Apr 15;185(8):842-50. doi: 10.1164/rccm.201107-1332OC. Epub 2012 Jan 26. PMID 22281833